CLINICAL TRIAL: NCT04833257
Title: Efficacy and Safety of of GP Chemotherapy Combined With Tislelizumab Neoadjuvant Therapy in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma: a Single-arm, Phase 2 Trial
Brief Title: Neoadjuvant Therapy of GP Chemotherapy Combined With Tislelizumab in Locoregionally Advanced NPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-FXY-484
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2021-04

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GP combine with Tislelizumab neoadjuvant therapy+CCRT (Experimental): Patients receive neoadjuvant therapy with gemcitabine(1000mg per square meter on day 1,8) , cisplatin (80mg per square meter on day 1) and tislelizumab(200mg) every three weeks for three cycles before radiotherapy, then followed by concurrent IMRT and cisplatin (100mg per square meter) concurrent every three weeks during radiotherapy (D1,D22,D43 of RT) .
  Interventions: Drug: GP combine with Tislelizumab neoadjuvant therapy+CCRT

INTERVENTIONS:
Drug: GP combine with Tislelizumab neoadjuvant therapy+CCRT — chemotherapy combine with anti-PD-1 targeted immunotherapy+concurrent chemotherapy

SUMMARY:
The purpose of this study is to explore the efficacy and safety of a combination of GP chemotherapy and tislelizumab in neoadjuvant therapy of locoregionally advanced nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
Platinum-based concurrent chemoradiotherapy is the standard of care for patients with locoregionally advanced nasopharyngeal carcinoma(NPC). Gemcitabine plus cisplatin(GP) has been demonstrated an effective chemotherapy regimen for NPC patients in previous studies. The results of GP combined with concurrent chemoradiotherapy in the treatment of locoregionally advanced nasopharyngeal carcinoma showed 10% of locoregionally advanced NPC patients had complete response after three cycles of GP neoadjuvant chemotherapy, and GP neoadjuvant chemotherapy added to chemoradiotherapy significantly improved recurrence-free survival (85.3% vs 76.5%) and overall survival (94.6% vs 90.3%) among locoregionally advanced NPC patients , as compared with chemoradiotherapy alone. Therefore, GP regimen has been established as the highest level of evidence-based neoadjuvant chemotherapy in the 2020 National Comprehensive Cancer Network (NCCN) guidelines. Recently, immune checkpoint inhibitors, such as anti-programmed cell death-1 (PD-1)monoclonal antibody has shown promising efficacy in the treatment of tumor patients. Clinical trials have shown objective response rates of 20.5%-34% in patients with recurrent or metastatic NPC patients receiving anti PD-1 monoclonal antibody immunotherapy including pembrolizumab, nivolumab, camrelizumab, and toripalimab. The current NCCN guidelines recommend anti PD-1 monoclonal antibody as a second-line treatment for recurrent or metastatic NPC. More and more evidence show that immunotherapy combined with chemotherapy has a synergistic effect in treating tumors. GP chemotherapy combined with anti PD-1 antibody has achieved the initial effect in NPC. Phase 1 trials have shown the combination of camrelizumab plus GP chemotherapy in recurrent or metastatic NPC led to a proportion of 91% patients achieving an objective response. Tislelizumab, approved by the National Medical Products Administration in China, is an anti-PD-1 monoclonal IgG4 antibody with higher affinity to PD-1 than pembrolizumab and nivolumab and was engineered to minimize binding to FcγR on macrophages in order to abrogate antibody-dependent phagocytosis, a mechanism of T-cell clearance and potential resistance to anti-PD-1 therapy. Multiple clinical trials have shown strong anti-neoplastic activity of tislelizumab in various tumors including NPC. Clinical trial has shown an objective response rates of 43% in patients with recurrent metastatic nasopharyngeal carcinoma treated with tirelizumab, which is superior to other anti PD-1 monoclonal antibodys. So we hypothesize that GP neoadjuvant chemotherapy combined with tislelizumab could further improve survival of patients with locaregionally advanced NPC. Based on this, this study aims to evaluate the efficacy and safety of gemcitabine plus cisplatin chemotherapy combined with tislelizumab neoadjuvant therapy, followed by cisplatin based concurrent chemoradiotherapy in the patients with locoregionally advanced nasopharyngeal carcinoma, to provide new evidence for individualized comprehensive treatment in NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation with Written informed consent.
2. Age ≥ 18 years and ≤ 70 years, male or non-pregnant female.
3. Histologically or cytologically confirmed with Nonkeratinizing carcinoma of the nasopharynx (differentiated or undifferentiated type, WHO II or III).
4. Original clinical staged as III-IVa (according to the 8th AJCC edition), Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
5. White blood cell count (WBC)≥4.0×109 /L, Hemoglobin ≥ 90g/L, Platelet count ≥100×109/L.
6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN),serum total bilirubin (TBIL) ≤2.0 times the upper limit of normal (ULN) .
7. Adequate renal function: creatinine clearance rate≥60 ml/min .

Exclusion Criteria:

1. Patients with recurrent or metastatic nasopharyngeal carcinoma.
2. Histologically or cytologically confirmed with keratinizing squamous cell carcinoma of the nasopharynx.
3. Prior therapy with Systemic chemotherapy.
4. Women in the period of pregnancy, lactation, or reproductive without effective contraceptive measures.
5. Seropositivity for human immunodeficiency virus (HIV).
6. Known history of other malignancies (except cured basal cell carcinoma or carcinoma in situ of the cervix).
7. Prior exposure to immune checkpoint inhibitors,including anti-PD-1, anti-PD-L1, anti-CTLA-4 antibodies.
8. Patients with immunodeficiency disease or a history of organ transplantation.
9. Received large doses of glucocorticoids, anticancer monoclonal antibodies, or other immunosuppressants within 4 weeks.
10. Patients with severe dysfunction of heart, liver, lung, kidney or marrow.
11. Patients with severe, uncontrolled disease or infections.
12. Received other research drugs or in other clinical trials at the same time.
13. Refuse or fail to sign the informed consent .
14. Patients with other treatment contraindications.
15. Patients with personality or mental disorders, incapacity or limited capacity for civil conduct.
16. Hepatitis B surface antigen (HBsAg) positive and peripheral blood HBV deoxyribonucleic acid (HBV DNA) ≥1000cps/ml.
17. Patients with positive HCV antibody test will only be enrolled in this study if the PCR test for HCV RNA is negative.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Complete Response | 9 weeks
  CR assessed by independent reviewers, according to the Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI). Disease response evaluated after the completion of the neoadjuvant therapy. Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) .

SECONDARY OUTCOMES:
Pathological Complete Response | 9 weeks
  Pathological complete response defined as the complete disappearance of the tumor cells in biopsy tissue of nasopharynx after neoadjuvant therapy .
Overall Survival(OS) | 2 years
  The OS was defined as the duration from the date of registration to the date of death from any cause or censored at the date of the last follow-up.
Progress-free survival(PFS) | 2 years
  Progress-free survival is calculated from the date of registration to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up
Locoregional failure-free survival(LRRFS) | 2 years
  The LRRFS is evaluated and calculated from the date of registration until the day of first locoregional relapse or until the date of the last follow-up visit.
Distant metastasis-free survival(DMFS) | 2 years
  The DMFS is evaluated and calculated from the date of registration until the day of first distant metastases or until the date of the last follow-up visit.
Incidence rate of adverse events (AEs) | 2 years
  Analysis of treatment-related AEs (trAEs) and immune-related AEs (irAEs) are evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria.
PD-L1 expression level of tumor cell | 2 years
tumor-infiltrating lymphocytes (TILs) | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Su LI, MD, Study Chair — GCP center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhang L, Huang Y, Hong S, Yang Y, Yu G, Jia J, Peng P, Wu X, Lin Q, Xi X, Peng J, Xu M, Chen D, Lu X, Wang R, Cao X, Chen X, Lin Z, Xiong J, Lin Q, Xie C, Li Z, Pan J, Li J, Wu S, Lian Y, Yang Q, Zhao C. Gemcitabine plus cisplatin versus fluorouracil plus cisplatin in recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2016 Oct 15;388(10054):1883-1892. doi: 10.1016/S0140-6736(16)31388-5. Epub 2016 Aug 23. PMID 27567279
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Zhang J, Fang W, Qin T, Yang Y, Hong S, Liang W, Ma Y, Zhao H, Huang Y, Xue C, Huang P, Hu Z, Zhao Y, Zhang L. Co-expression of PD-1 and PD-L1 predicts poor outcome in nasopharyngeal carcinoma. Med Oncol. 2015 Mar;32(3):86. doi: 10.1007/s12032-015-0501-6. Epub 2015 Feb 22. PMID 25702326
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Background] Economopoulou P, Kotsantis I, Psyrri A. The promise of immunotherapy in head and neck squamous cell carcinoma: combinatorial immunotherapy approaches. ESMO Open. 2017 Feb 13;1(6):e000122. doi: 10.1136/esmoopen-2016-000122. eCollection 2016. PMID 28848660
- [Background] Desai J, Deva S, Lee JS, Lin CC, Yen CJ, Chao Y, Keam B, Jameson M, Hou MM, Kang YK, Markman B, Lu CH, Rau KM, Lee KH, Horvath L, Friedlander M, Hill A, Sandhu S, Barlow P, Wu CY, Zhang Y, Liang L, Wu J, Paton V, Millward M. Phase IA/IB study of single-agent tislelizumab, an investigational anti-PD-1 antibody, in solid tumors. J Immunother Cancer. 2020 Jun;8(1):e000453. doi: 10.1136/jitc-2019-000453. PMID 32540858
- [Background] Shen L, Guo J, Zhang Q, Pan H, Yuan Y, Bai Y, Liu T, Zhou Q, Zhao J, Shu Y, Huang X, Wang S, Wang J, Zhou A, Ye D, Sun T, Gao Y, Yang S, Wang Z, Li J, Wu YL. Tislelizumab in Chinese patients with advanced solid tumors: an open-label, non-comparative, phase 1/2 study. J Immunother Cancer. 2020 Jun;8(1):e000437. doi: 10.1136/jitc-2019-000437. PMID 32561638